CLINICAL TRIAL: NCT05483725
Title: Assessment of Association Between 3rd Dose of mRNA Vaccine and Risk of SARS-CoV-2 Infection in Kidney Transplant Recipients, Safety and Immunogenicity Assessment.
Brief Title: Immunological Safety and Effectiveness of the First Booster Dose of mRNA Vaccines Against COVID-19 in Kidney Transplant Recipients.
Status: Active, not recruiting | Type: Observational
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Prof. Ondřej Viklický, M.D., Ph.D., Head of the Transplant Center, Head of the Department of Nephrology, Principle Investigator, Clinical Professor, Institute for Clinical and Experimental Medicine
Other Study IDs: G-21-71
Record Dates: First submitted 2022-07-31; First posted 2022-08-02 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Kidney Diseases; Kidney Transplant; Complications; COVID-19; Vaccine Adverse Reaction; Rejection Acute Renal; Rejection Chronic Renal
Keywords: kidney transplantation; COVID-19; mRNA vaccine; vaccine safety; alloreactivity
MeSH Terms: conditions — Kidney Diseases; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples, four 5ml vials of blood, taken on day of booster dose and 3 months later.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- First booster dose group
  Interventions: Biological: Booster dose of mRNA vaccine

INTERVENTIONS:
Biological: Booster dose of mRNA vaccine — Administration of SARS-CoV-2 mRNA vaccine.

SUMMARY:
Prospective observational trial to assess immunological safety (anti-HLA antibodies, donor-derived cell-free DNA) and immunological effectiveness (anti-SARS-CoV-2 IgG) of the first booster dose of SARS-CoV-2 mRNA vaccines in kidney transplant recipients at least one year from transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipients followed at Institute for Clinical and Experimental Medicine (IKEM)
* vaccinated with 2 doses of mRNA vaccine (BNT-162b2 or mRNA-1273)
* immunosuppressive regimen includes or does not include mycophenolic acid or mycophenolate mofetil
* COVID naive

Exclusion Criteria:

* age < 18 years
* pregnant women, breastfeeding women
* unable/unwilling to give informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients, vaccinated with 2 doses of mRNA vaccines against COVID, scheduled for the first booster dose.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2024-12-04 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Immunological safety - anti-HLA antibodies | Comparison of anti-HLA single antigen bead assays at booster dose and three months later.
  Emergence of de novo anti-HLA/donor specific antibodies, increase of preformed anti-HLA/donor specific antibodies above 50% of pre-booster level.
Immunological safety - donor-derived cell-free DNA | Comparison of dd-cfDNA assays at booster dose and three months later.
  Elevation of dd-cfDNA above 1% threshold

SECONDARY OUTCOMES:
Immunological effectiveness - anti-SARS-CoV-2 antibodies | Comparison of anti-SARS-CoV-2 IgG assays at booster dose and three months later.
  Emergence or increase of anti-SARS-CoV-2 IgG.

CONTACTS AND LOCATIONS:
Overall Officials: Ondrej Viklicky, MD, PhD, Principal Investigator — Head of Department of Nephrology
Locations (1):
- Institute for Clinical and Experimental Medicine, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Petr V, Zahradka I, Modos I, Roder M, Fialova M, Machkova J, Kabrtova K, Hruba P, Magicova M, Slavcev A, Striz I, Viklicky O. Safety and Immunogenicity of SARS-CoV-2 mRNA Vaccine Booster Doses in Kidney Transplant Recipients: Results of a 12-mo Follow-up From a Prospective Observational Study. Transplant Direct. 2024 May 17;10(6):e1645. doi: 10.1097/TXD.0000000000001645. eCollection 2024 Jun. PMID 38769974
- [Derived] Petr V, Zahradka I, Modos I, Roder M, Prewett A, Fialova M, Machkova J, Hruba P, Magicova M, Slavcev A, Striz I, Viklicky O. First Booster of SARS-COV-2 mRNA Vaccine Is Not Associated With Alloimmunization and Subclinical Injury of Kidney Allograft. Transplantation. 2023 Feb 1;107(2):e62-e64. doi: 10.1097/TP.0000000000004421. Epub 2022 Oct 29. No abstract available. PMID 36314999